CLINICAL TRIAL: NCT04058964
Title: A Pilot Study to Assess the Efficacy and Safety Effects of Pembrolizumab and PEGPH20 (Pegvorhyaluronidase Alfa) in Patients With Metastatic Pancreatic Cancer
Brief Title: Pembrolizumab and PEGPH20 in Treating Patients With Metastatic Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn by supporter
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0342; NCI-2019-04856 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0342 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — PEGPH20; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, PEGPH20) (Experimental): Patients receive pembrolizumab IV over 10 minutes on day 1 and pegylated recombinant human hyaluronidase PH20 SC on days 1, 8, and 15. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pegylated Recombinant Human Hyaluronidase PH20; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pegylated Recombinant Human Hyaluronidase PH20 — Given SC
  Other Names: PEGPH20; Pegylated Recombinant Human PH20; Pegylated rHuPH20; PH20
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and PEGPH20 work in treating patients with pancreatic cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. PEGPH20 is an enzyme that breaks down hyaluronic acid coating tumor cells which may inhibit growth of tumor cells. Giving pembrolizumab and PEGPH20 may work better in treating patients with pancreatic cancer compared to pembrolizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the progression free survival duration of patients treated with the combination of pegylated recombinant human hyaluronidase PH20 (PEGPH20) and pembrolizumab.

SECONDARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of PEGPH20 and pembrolizumab.

EXPLORATORY OBJECTIVES:

I. To evaluate objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) and Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria, duration of response (DOR), disease control rate (DCR), time to progression (TTP) and progression-free survival (PFS) per RECIST and iRECIST as assessed by M.D. Anderson investigators and overall survival (OS) of the combination of pembrolizumab and PEGPH20.

II. To explore the association between PD-L1 expression by immunohistochemistry (IHC), shed PD-L1 level, hyaluronan (HA) levels, somatic gene expression profiling and antitumor efficacy of the combination of pembrolizumab and PEGPH20 based on RECIST 1.1 as well as OS.

III. To explore the relationship between genomic variation and response to study treatment.

IV. To examine the effect of pembrolizumab and PEGPH20 on immune cell infiltration into tumor.

V. To explore the effect of PEGPH20 on serum HA levels, and to compare changes in serum HA with clinical efficacy.

VI. To determine the impact of the combination of pembrolizumab and PEGPH20 on circulating immune cells.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 10 minutes on day 1 and pegylated recombinant human hyaluronidase PH20 subcutaneously (SC) on days 1, 8, and 15. Cycles repeat every 21 days for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 9 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma based on pathology report
* Be willing and able to provide written informed consent for the trial. The subject may also provide consent for Future Biomedical Research. However, the subject may participate in the main trial without participating in Future Biomedical Research.
* Have at least one measurable lesion and one lesion available for biopsy (not the primary pancreatic lesion) based on RECIST 1.1. Target lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Have had prior treatment with first-line therapy for metastatic disease for at least 4 months, and have had a radiologic response or stable disease at the most recent imaging. Adjuvant therapy for resected disease will not count as first-line therapy. Therapies that are derivative of others (e.g. fluorouracil/leucovorin calcium/oxaliplatin [FOLFOX] vis-a-vis fuorouracil/irinotecan/leucovorin/oxaliplatin [FOLFIRINOX]) will be counted as a single line of treatment for the purpose of determining the number of prior therapies
* Be willing to undergo a core biopsy or excisional biopsy of tumor from a metastatic site. Note that the biopsy itself will be done only after the patient has been found to meet all other inclusion/exclusion criteria and the patient is otherwise prepared to start therapy
* Be willing to provide (and have available) archival tissue from a surgical or biopsy specimen obtained PRIOR to the most recent chemotherapy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Demonstrate adequate organ function. Specimens must be collected within 10 days prior to the start of trial treatment
* Female subjects of childbearing potential must have a negative urine or serum pregnancy test at screening (prior to biopsy) and again within 24 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Male and female subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of trial therapy through 120 days after the last dose of trial therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject. Acceptable methods of contraception are as follows:

  * Single method (1 of the following is acceptable): intrauterine device (IUD), vasectomy of a female subject's male partner, contraceptive rod implanted into the skin
  * Combination method (requires use of 2 of the following): diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide), cervical cap with spermicide (nulliparous women only), contraceptive sponge (nulliparous women only), male condom or female condom (cannot be used together), hormonal contraceptive: oral contraceptive pill (estrogen/ progestin pill or progestin-only pill), contraceptive skin patch, vaginal contraceptive ring, or subcutaneous (SC) contraceptive injection

Exclusion Criteria:

* Has pancreatic tumor other than adenocarcinoma, including: acinar cell carcinoma, pancreaticoblastoma, malignant cystic neoplasms, endocrine neoplasms, squamous cell carcinoma, ampulla of Vater, periampullary, duodenal, or common bile duct malignancies
* Has had more than one line of systemic chemotherapy for metastatic disease
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has had prior treatment with PEGPH20
* Has received prior systemic anti-cancer therapy that includes investigational agents within 2 weeks prior to treatment
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Had a solid organ or hematologic transplant
* Has active autoimmune disease that has required systemic treatment in past 3 months (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Patients with autoimmune colitis (eg Crohn's disease) will be excluded. Any relevant diseases not listed here are to be discussed with the study supporters. Replacement hormone therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has a diagnosed additional malignancy within 1 year prior to first dose of study treatment, with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected tumors of low invasive potential (e.g. in situ cervical and/or breast cancers)
* Has a history of central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a history of (non-infectious) pneumonitis that required oral or IV steroids or currently has pneumonitis
* Has an active infection requiring systemic therapy
* Chronic use of steroids for pain or emesis management
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has received prior immunotherapy including anti-PD-1, anti-PD-L1, or anti-PD-L2 agents, or with an agent directed to another stimulatory or co-inhibitory T cell receptor (eg, CTLA-4, OX-40, CD137), or has previously participated in Merck pembrolizumab or PEGPH20 clinical trials
* Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies) (HIV testing is required during screening)
* Has a history of the following liver diseases: hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive), hepatitis C (defined as detectable hepatitis C virus [HCV] ribonucleic acid [RNA]), primary biliary cholangitis, primary sclerosing cholangitis, history of immune mediated cholangitis. Of note, patients with a history of bacterial cholangitis are eligible if the infection has been fully resolved prior to the screening visit. An exception is made for hepatitis C patients who have undergone treatment and who have negative serologic testing for at least one year
* Has received a live vaccine within 30 days prior to the first dose of trial drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist) are live attenuated vaccines and are not allowed
* Has a known history of active TB (Bacillus tuberculosis)
* Is unable to tolerate a contrast enhanced computed tomography (CT) or magnetic resonance imaging (MRI) for staging/restaging purposes
* Has not recovered (i.e., grade 1 or at baseline) from adverse events (AEs) due to chemotherapy (neuropathy and alopecia are excluded)
* Has clinical evidence of a deep vein thrombosis (DVT), pulmonary embolism (PE), or other known thrombotic event present during the screening period. Of note - this does not apply to splanchnic vein (eg portal / superior mesenteric vein) thrombosis that, in the opinion of the primary investigator, are primarily associated with the anatomic location of the underlying disease
* Requires Megace (medroxyprogesterone acetate)
* In the estimation of the treating physician or primary investigator, have had a clinical deterioration of their ECOG performance within the month prior to enrollment
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has unstable angina, new onset angina within the last 3 months, myocardial infarction within the last 6 months, and current congestive heart failure New York Heart Association class III or higher. Additionally, subjects with myocardial infarction or atrial fibrillation within the past 12 months are excluded
* Has a history of a cerebrovascular accident or transient ischemic attack
* Known clinically significant pre-existing carotid artery disease
* Has a history of active bleeding requiring transfusion within a 3 month period prior to screening
* Known allergy/intolerance to hyaluronidase or dexamethasone
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients
* Contraindication to heparin or non-steroidal anti-inflammatory drugs (NSAIDs)
* Known cases of drug-induced hepatobiliary toxicities (other than a radiological finding of fatty liver)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Up to 1 year
  Descriptive statistics including with 90% confidence interval will be computed.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post treatment
  Descriptive statistics including with 90% confidence interval will be computed.

OTHER OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  ORR will be evaluated per Response Evaluation Criteria in Solid Tumors (RECIST) and Immune-Modified Response Evaluation Criteria in Solid Tumors (iRECIST) criteria. Descriptive statistics including with 90% confidence interval will be computed.
Duration of response (DOR) | Up to 1 year
  DOR will be evaluated per RECIST and iRECIST. Descriptive statistics including with 90% confidence interval will be computed.
Disease control rate (DCR) | Up to 1 year
  DCR will be evaluated per RECIST and iRECIST. Descriptive statistics including with 90% confidence interval will be computed.
Time to progression (TTP) | Up to 1 year
  TTP will be evaluated per RECIST and iRECIST. Descriptive statistics including with 90% confidence interval will be computed.
PFS | Up to 1 year
  PFS will be evaluated per RECIST and iRECIST. Descriptive statistics including with 90% confidence interval will be computed.
Overall survival | Up to 1 year
  Descriptive statistics including with 90% confidence interval will be computed.

CONTACTS AND LOCATIONS:
Overall Officials: David R Fogelman, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org